CLINICAL TRIAL: NCT02754336
Title: Working Memory Training and Neurofeedback for Children With ADHD, a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SUS_ID2012/439
Record Dates: First submitted 2015-11-22; First posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Neurofeedback

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cogmed Robomemo, working memory training (Active Comparator): Robomemo working memory training, 25 sessions with 8 verbal and non-verbal tasks per session.
  Interventions: Behavioral: Cogmed Robomemo, working memory training
- Othmer, neurofeedback (Active Comparator): Othmer method neurofeedback, 25 sessions a 30 minutes.
  Interventions: Behavioral: Othmer, neurofeedback

INTERVENTIONS:
Behavioral: Cogmed Robomemo, working memory training
  Arms: Cogmed Robomemo, working memory training
Behavioral: Othmer, neurofeedback
  Arms: Othmer, neurofeedback

SUMMARY:
This pilot study compares the effect of working memory training and neurofeedback in non-medicated children age 7 to 13 years with ADHD. Half of the participants will receive working memory training, while the other half will receive neurofeedback.

ELIGIBILITY:
Inclusion Criteria:

* ADHD/ADD

Exclusion Criteria:

* Positive effect of metylphenidate

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2014-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Neuropsychological tests | 3-4 weeks after last training session
  Subtests from the NEPSY-II test battery

SECONDARY OUTCOMES:
Quantum EEG | 3-4 weeks after last training session
  Electroencephalography (EEG) is the measurement of electrical patterns at the surface of the scalp which reflect cortical activity, and are commonly referred to as "brainwaves". Quantitative EEG (qEEG) is the analysis of the digitized EEG, and in lay terms this sometimes is also called "Brain Mapping"
Questionaires | 3-4 weeks after last training session
  5-15 (FTF) Parent Questionaire For Evaluation of Development and Behavior of 5 to 15-year-old children. Behavior Rating Inventory of Executive Function (BRIEF)

CONTACTS AND LOCATIONS:
Overall Officials: Harald Beneventi, PhD, Principal Investigator — Helse Stavanger HF
Locations (1):
- Stavanger University Hospital, Stavanger, Norway

IPD SHARING:
Plan to Share IPD: No